CLINICAL TRIAL: NCT03755908
Title: Sensitivity of Forced Oscillation Technique (FOT) in Children With Asthma and Normal Spirometry
Brief Title: Sensitivity of Forced Oscillation Technique in Children With Asthma and Normal Spirometry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0384-18-RMB-CTIL
Record Dates: First submitted 2018-10-16; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Asthma in Children
Keywords: Forced oscillation technique; Airway obstruction; Asthma
MeSH Terms: conditions — Airway Obstruction; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- asthmatic children: Children with the diagnosis of asthma and normal spirometry results. Each subject will undergo evaluation including: asthma control questionnaire, spirometry, FOT and Fractional exhaled nitric oxide (FeNO).
  Interventions: Device: Forced oscillation technique (FOT)

INTERVENTIONS:
Device: Forced oscillation technique (FOT) — FOT will be measured using the TremoFlo C-100 Airwave Oscillometry System (Thorasys , Montreal, Quebec, Canada). R5, R20, R5-20 (resistances in the reported frequency), X5 (reactance in 5hz) and Ax5 (reactance area in 5hz) will be reported.

SUMMARY:
Exhibiting variable airway obstruction is a key factor in the diagnosis of asthma but too often it is undetected by spirometry.

Study hypothesis: The forced oscillation technique (FOT) will show airway obstruction in asthmatic children with normal spirometry pointing out its advantage in measuring AW obstruction in this population.

We will conduct a prospective observational study in 6-18 years old children with the diagnosis of asthma and a normal spirometry results.

Each subject will undergo evaluation including: asthma control questionnaire, spirometry, FOT and Fractional exhaled nitric oxide (FeNO) to assess the sensitivity of FOT in diagnosing airway obstruction in this circumstances.

DETAILED DESCRIPTION:
Background: Asthma diagnosis and control are based on history of recurrent typical symptoms and variable airflow obstruction by by measuring maximal expiratory flows with spirometry. However, in many children with asthma spirometry can be normal. The forced oscillation technique (FOT) is a simple, noninvasive technique performed during tidal breathing that is relatively easy to apply.

The objective of this study is to assess the sensitivity of FOT in children with asthma and normal spirometry.

Study design: this will be a prospective observational study. Population: 6-18 years old children visiting the pediatric pulmonary clinic at the investigators institution with the diagnosis of asthma and normal spirometry results (FEV1 & FEV1/FVC >80% and FEF25-75>65%) either on treatment or before treatment.

Study protocol:

After obtaining written informed consent, participants will fill asthma control questionnaires. Family history and risk factors for asthma will be reviewed. Data on blood eosinophils and skin prick test for allergy will be collected from the medical files. Medication (controller and reliever) will be also documented.

FOT will be measured using the TremoFlo C-100 Airwave Oscillometry System (Thorasys , Montreal, Quebec, Canada). R5, R20, R5-20 (resistances at the reported frequency), X5 (reactance at 5hz), AX5 (reactance area at 5hz), Fres (resonance frequency) will be reported.

Fractional exhaled nitric oxide (FeNO) will be measured using the single breath exhalation technique.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Must be able to perform spirometry and FOT tests
* Normal spirometry results (FEV1 & FEV1/FVC >80% and FEF25-75>65%)

Exclusion Criteria:

* Chronic lung disease other than asthma
* Severe chronic medical condition such as heart failure, neuromuscular disease etc.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with the diagnosis of asthma and a normal spirometry results
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
R5 | One year
  Resistances at the frequency of 5 hertz in kilopascal per liter per second
R20 | One year
  Resistances at the frequency of 20 hertz in kilopascal per liter per second
R5-R20 | One year
  The difference between R5 to R20 in kilopascal per liter per second
Xrs 5 | One year
  Reactance at the frequency of 5 hertz in kilopascal per liter

SECONDARY OUTCOMES:
FeNO | One year
  Fractional exhaled Nitric Oxide (parts per billion)

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Principal Investigator — Rambam Medical Center, Haifa, Israel
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No